CLINICAL TRIAL: NCT03540407
Title: Efficacy of the Oncoxin-Viusid® Oral Solution in Reducing the Adverse Reactions of Chemotherapy and Radiotherapy in Patients Diagnosed With Cervical Cancer and Endometrial Adenocarcinoma.
Brief Title: Evaluation of Oncoxin-Viusid® in Cervical Cancer and Endometrial Adenocarcinoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-3
Record Dates: First submitted 2018-05-03; First posted 2018-05-30 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Cervical Carcinoma Stage II; Cervical Carcinoma Stage III; Cervical Carcinoma Stage IV; Endometrial Adenocarcinoma Stage II; Endometrial Adenocarcinoma Stage III; Endometrial Adenocarcinoma Stage IV
Keywords: Cervical carcinoma; Endometrial adenocarcinoma; Oncoxin-Viusid; Nutritional supplement; Antioxidant
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oncoxin-Viusid® (Experimental): will receive the Oncoxin-Viusid® (oral solution) concomitant to the onco-specific treatment.
  Interventions: Dietary Supplement: Oncoxin-Viusid®
- Placebo (Placebo Comparator): will receive a Placebo concomitant to the onco-specific treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oncoxin-Viusid® — Administration of the Oncoxin-Viusid® oral solution 25 mL three times a day during the concurrent Radiotherapy and Chemotherapy treatment and up to 3 weeks after the end of the onco-specific treatment
  Arms: Oncoxin-Viusid®
Dietary Supplement: Placebo — Administration of the Oncoxin-Viusid® oral solution placebo 25 ml three times a day during the concurrent Radiotherapy and Chemotherapy treatment and up to 3 weeks after the end of the onco-specific treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of oral solution Oncoxin-Viusid in the reduction of acute toxicity of Radiotherapy (RTP) and Chemotherapy (QTP) in patients with histological diagnosis of cervical cancer and endometrial adenocarcinoma. This is a phase II, prospective, randomized and double blind clinical trial, which will include 66 patients assigned to 2 treatment arms: 33 patients will receive conventional treatment, plus a placebo of the nutritional supplement and another 33 patients will receive along with the conventional treatment the Oncoxin-Viusid nutritional supplement produced by the Catalysis Laboratories of Spain. Patients will receive oral treatment throughout the onco-specific treatment and up to 3 weeks after completion.

DETAILED DESCRIPTION:
Patients will be evaluated clinically and hematological at the beginning of the treatment, before each cycle of treatment with QTP / RTP, at month, two and three months after the end of the treatment with follow-up every three months for 1 year. The self-perceived quality of life related to health will be assessed by means of the EORTC questionnaires (QLQ-C30 and the specific questionnaire QLQ-CX24) at the beginning and a year after completing the treatment. The toxicity to the research product will be described according to Common Criteria of Terminology for the Report of Adverse Events (CTCAE version 4) and the tolerance to onco-specific treatment. It is expected that with the joint administration of the research product, the patients will have a better tolerance to the treatment of QTP / RTP with a decrease of the interruptions by toxicity in 25% and will preserve a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmation of cervical cancer and adenocarcinoma of the endometrium that are treated with chemotherapy and ionizing radiation.
* Patient with age equal to or greater than 18 years and up to 80 years.
* Patients who do not present decompensated concurrent diseases at the time of diagnosis that prevent or contraindicate the application of treatment with chemo-radiotherapy.
* Informed consent to participate in the investigation.
* Patients with an ECOG <or equal to 3.

Exclusion Criteria:

* Patients with a history of renal failure that contraindicates the administration of cisplatin.
* Concomitant diseases unbalanced at the time of diagnosis or during the application of treatment.
* Patients with an ECOG> 3.
* Pregnant or lactating women.
* Patients who are receiving another research product.
* Patients who do not show consent to participate in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women
Enrollment: 66 (Estimated)
Dates: Start 2015-01-07 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Toxicity of chemotherapy and radiotherapy in patients diagnosed with cervical cancer and endometrium adenocarcinoma. | 3 months
  Patients diagnosed with cervical cancer and adenocarcinoma of the endometrium usually have varying degrees of malnutrition and immunodeficiencies; they are carriers of oncogenic virus infections, and present deterioration of their general state, depression-anxiety and socio-economic dysfunctions. Oncospecific treatment's toxicity is measured according to Common Criteria of Terminology for the Report of Adverse Events (CTCAE version 4).

SECONDARY OUTCOMES:
quality of life | 3 months
  Self-perceived quality of life related to health through the EORTC test QLQ-C30 at the beginning and at the end of the treatment.
Reduce hospital costs | 3 months
  Reduce hospital costs by being unnecessary or decreasing, the use of concomitant support treatments that counteract the adverse effects caused by these, hospitalization for the treatment of complications secondary to the treatment of QTP / RTP and the use of antibiotics in cases of neutropenia / leukopenia and sepsis added, very frequent in these patients.
Quality of life | 3 months
  Self-perceived quality of life related to health through the EORTC test QLQ-CX24 at the beginning and at the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Raiza Ruiz Llorente, Dr., Principal Investigator — Ramón González Coro Hospital
Locations (1):
- Ramón González Coro Hospital, La Habana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR